CLINICAL TRIAL: NCT02183311
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses (1 to 10 mg) and Multiple Rising Oral Doses (2.5 to 10 mg Once Daily for 12 Days) of BI 1356 BS in Healthy Male Volunteers (a Randomised, Double-blind, Placebo Controlled Within Dose Groups Clinical Trial)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses and Multiple Rising Oral Doses of BI 1356 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.11
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- BI 1356 BS - single rising dose (Experimental)
  Interventions: Drug: BI 1356 BS - single rising dose
- BI 1356 BS - multiple rising dose (Experimental)
  Interventions: Drug: BI 1356 BS - multiple rising dose
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356 BS - single rising dose
  Arms: BI 1356 BS - single rising dose
Drug: BI 1356 BS - multiple rising dose
  Arms: BI 1356 BS - multiple rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to examine the safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 1356 BS administered to healthy male volunteers at single rising oral doses (1 mg, 2.5 mg, 5 mg, and 10 mg) and at multiple rising oral doses (2.5 mg, 5 mg, and 10 mg once daily for 12 days)

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy male volunteers who meet the criteria below: Persons without clinically remarkable findings or clinically evident complications based on their concurrent illness, past medical history, physical examination, vital signs (blood pressure (BP), pulse rate (PR), and body temperature), 12-lead Electrocardiogram (ECG), and laboratory test results
* Persons who are 20 or older and 35 or younger
* Persons with a BMI 17.6 kg/m2 or more and 29.9 kg/m2 or less
* Persons who are willing to participate in this trial before study initiation and who give their written consent in accordance with GCP (Good Clinical Practice, MHW Ordinance No. 28 dated March 27, 1997)

Exclusion Criteria:

* Persons who deviate from the norm and who show clinical findings (BP, PR, and ECG) on consultation
* Persons with any clinically relevant complications
* Persons with gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immune, or hormonal disorders
* Persons with central nervous system disorders (e.g., epilepsy), mental disorders, or neurological disorders
* Persons with a history of significant orthostatic hypotension, syncopal attacks, or blackouts
* Persons with chronic infection or severe acute infection
* Persons with a history of severe allergy/hypersensitivity including allergies to drugs and inactive ingredients
* Persons who will have received a drug with a long half-life (more than 24 hours) within the month before treatment in this trial, within a period 10 times longer than the half-life of each drug, or during the study
* Persons who will have received a drug that may theoretically affect the study results based on the information obtained at the time of preparation of the protocol within the 10 days before treatment or during the study
* Persons who will have participated in another trial of an investigational drug within the 4 months before treatment or during the study
* Smokers (who smoke more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Persons who cannot abstain from smoking throughout the study
* Persons who undoubtedly abuse alcohol
* Persons who abuse drugs
* Persons who donate blood of 100 mL or more within the 4 weeks before treatment
* Persons who perform rigorous exercise (within the week before treatment or during the study)
* Persons with any laboratory test result outside the reference range and for whom the result is considered a clinically relevant change
* Persons who cannot obey the dieting rules of the trial site
* Persons with any ECG value outside the reference range and who are of clinical importance. Examples include, but are not limited to, QRS interval>120 ms

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-06; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Screening, up to 28 days
Number of patients with clinically significant changes in Vital signs (blood pressure [BP], pulse rate [PR]) | Screening, up to 28 days
Number of patients with abnormal findings in 12-lead electrocardiogram (ECG) | Screening, up to 28 days
Number of patients with abnormal changes in laboratory parameters | Screening, up to 28 days
Number of patients with adverse events | up to 49 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 192 h (single dose), up to 456 h (multiple dose)
tmax (time from dosing to maximum measured concentration) | up to 192 h (single dose), up to 456 h (multiple dose)
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 192 h (single dose), up to 456 h (multiple dose)
%AUCtz-∞ (the percentage of the AUCtz-∞ that is obtained by extrapolation) | up to 192 h (single dose), up to 456 h (multiple dose)
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable analyte plasma concentration) | up to 192 h (single dose), up to 456 h (multiple dose)
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval from the time point t1 to the time point t2) | up to 192 h (single dose), up to 456 h (multiple dose)
λz (terminal rate constant in plasma) | up to 192 h (single dose), up to 456 h (multiple dose)
t1/2 (terminal half-life of the analyte in plasma) | up to 192 h (single dose), up to 456 h (multiple dose)
MRTpo (mean residence time of the analyte in the body) | up to 192 h (single dose), up to 456 h (multiple dose)
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | up to 192 h (single dose), up to 456 h (multiple dose)
Vz/F (apparent volume of distribution during the terminal phase λz following extravascular administration) | up to 192 h (single dose), up to 456 h (multiple dose)
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to the time point t2) | up to 192 h (single dose), up to 456 h (multiple dose)
fet1-t2 (fraction of analyte eliminated in urine from the time point t1 to the time point t2) | up to 192 h (single dose), up to 456 h (multiple dose)
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 192 h (single dose), up to 456 h (multiple dose)
CLR,0-24,1 (renal clearance of the analyte from 0 until 24 hours after administration of the first dose) | up to 192 h (single dose), up to 456 h (multiple dose)
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 192 h (single dose), up to 456 h (multiple dose)
Cavg (average concentration of the analyte in plasma at steady state) | up to 192 h (single dose), up to 456 h (multiple dose)
Cpre (predose concentration of the analyte in plasma) | up to 192 h (single dose), up to 456 h (multiple dose)
RA,Cmax based on Cmax | up to 192 h (single dose), up to 456 h (multiple dose)
RA,AUC based on AUCτ | up to 192 h (single dose), up to 456 h (multiple dose)
Emin (minimum Dipeptidyl-Peptidase IV (DPP-IV) activity | up to 192 h (single dose), up to 456 h (multiple dose)
tmin (time to reach minimum DPP-IV activity) | up to 192 h (single dose), up to 456 h (multiple dose)
E24 (DPP-IV activity 24 hours after administration of single dose administration and the first dose of multiple dose administration) | up to 192 h (single dose), up to 456 h (multiple dose)